CLINICAL TRIAL: NCT02756923
Title: Regulation of Stem Spermatogonia in the Mature Testis
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1202012193; 1P50HD096723-01A1 (NIH)
Record Dates: First submitted 2016-04-13; First posted 2016-04-29 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Male Infertility
Keywords: Male Infertility; Spermatogonial stem cell
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Testicular tissue, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigative trial to evaluate the role of a glial cell lined derived neurotrophic factor (GDNF) in regulation of spermatogonial renewal and testicular function. Goal of the trial is to provide greater information on the mechanisms that effect stem spermatogonial maintenance renewal and proliferation in its relation to male infertility.

DETAILED DESCRIPTION:
An essential requirement for sustaining male fertility is maintaining an adequate number of stem spermatogonia, the foundation of spermatogenesis. To achieve this, when the stem cells divide, some progeny must remain stem spermatogonia while other progeny differentiate. It is obvious that the correct balance between self-renewing replication and differentiation of stem spermatogonia is crucial to male fertility, and there is a indirect evidence that GDNF plays an important role in maintaining this balance in the normal mature testis. However, almost nothing is known about the in vivo regulation of this balance in the mature organ, of the specific function of GDNF in the adult testis, or if physiological changes in GDNF expression significantly affect the replication or differentiation of the stem cells. To address these critical issues, a unique mouse model that allows GDNF signaling to the stem spermatogonia to be specifically and reversibly inhibited in vivo by an ATP antagonist. With this model, the first direct evidence that GDNF is required for maintaining the stem spermatogonial pool in a normal mature testis. Additionally, the investigators have shown that when inhibition of GDNF signaling is reversed, the stem cells begin to rebuild the stem cell pool. Importantly, our data demonstrate that some stem spermatogonia are lost when GDNF signaling is inhibited for as little as 2 days, while other stem cells survive for up to 11 days. This suggests that factors intrinsic or extrinsic to the stem cells modulate the response to GDNF. Using this new mouse model the mechanisms responsible for the loss of stem spermatogonia proliferation and regeneration will be investigated along with GDNF signaling and inhibition. At the end of all of this these studies will be done on waste tissue obtained from normal men and men with infertility who otherwise have testicular surgery for therapeutic purposes.

ELIGIBILITY:
Inclusion Criteria:

* undergoing testicular biopsy at Weill Cornell Medicine/New York Presbyterian

Exclusion Criteria:

* females and any males outside of the age parameter of 18-75 years old

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy males undergoing testicular biopsy by any urologic surgeon at Weill Cornell Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2012-04; Primary Completion 2019-11-07 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Levels of glial cell line derived neurotrophic factor (GDNF) in normal testis compared to abnormal testicular tissue obtained from infertile patients | five years
  Levels of glial cell line derived neurotrophic factor (GDNF) in normal testis compared to abnormal testicular tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Schlegel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh D, Paduch DA, Schlegel PN, Orwig KE, Mielnik A, Bolyakov A, Wright WW. The production of glial cell line-derived neurotrophic factor by human sertoli cells is substantially reduced in sertoli cell-only testes. Hum Reprod. 2017 May 1;32(5):1108-1117. doi: 10.1093/humrep/dex061. PMID 28369535
- [Result] Paduch DA, Hilz S, Grimson A, Schlegel PN, Jedlicka AE, Wright WW. Aberrant gene expression by Sertoli cells in infertile men with Sertoli cell-only syndrome. PLoS One. 2019 May 9;14(5):e0216586. doi: 10.1371/journal.pone.0216586. eCollection 2019. PMID 31071133